CLINICAL TRIAL: NCT04028622
Title: Validation of Telemedicine Pre-anesthesia Consultation in Low-risk Anesthetic Patients Undergoing Ambulatory Surgery
Acronym: ANESTHADOM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The insufficient development of connection networks limit the teleconsultation deployment in the Grenoble metropolitan area
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Agence Régionale de Santé Rhône-Alpes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 38RC17.217
Record Dates: First submitted 2019-03-18; First posted 2019-07-22 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Outpatient Surgery; Telemedicine
Keywords: ambulatory; anesthesia; consultation; telemedicine
MeSH Terms: interventions — thiazole-4-carboxamide adenine dinucleotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCAD (telemedicine anesthesia consultation) (Experimental): Patients having a telemedicine anesthesia consultation
  Interventions: Other: TCAD (telemedicine anesthesia consultation)

INTERVENTIONS:
Other: TCAD (telemedicine anesthesia consultation) — Patients in the TCAD (telemedicine anesthesia consultation) group, arrange their bookings on a website and realise their anesthesia consultation from a platform from home

SUMMARY:
The purpose of this study is to validate the teleconsultation of anesthesia in anesthetic low risk patients and undergoing outpatient surgery.

DETAILED DESCRIPTION:
Anesthesia consultation is a necessary and obligatory step in the process of anesthesia. Telemedicine anesthesia consultation (TCAD) experiments have been successfully conducted in the United States, demonstrating the technical feasibility and medical relevance of the approach. In partnership with the Rhône-Alpes Regional Health Agency, an Telemedicine anesthesia consultation will be set up at the University Hospital Grenoble for low-risk anesthetic and surgical patients via a telemedicine platform accessible to patients' homes. Avoiding transport, unclog consultations in hospitals, and avoiding absences from work for traditional consultations are some of the advantages of this new method of consultation. This project involves assessing the feasibility, safety, and costs associated with home anesthesia teleconsultation for patients requiring outpatient surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for ambulatory surgery with anesthesia procedures
* Patients with American Society of Anesthesiologists score 1 or 2.
* Patients with visual and auditory acuity, language proficiency.
* Non-urgent surgery
* Affiliation to the French Social Security

Exclusion Criteria:

* patient with American Society of Anesthesiologists score 2 and complex treatments
* Complex surgical procedure
* Patient taking anticoagulant and / or antiplatelet treatments
* Patient having a serious problem during a previous surgery
* Pregnant woman
* Patient under guardianship or deprivation of liberty by judicial decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Validation of anesthesia teleconsultation in low-risk anesthetic patients undergoing outpatient surgery | 24 hours post surgery
  Patients rate with performed surgery following a successful telemedicine anesthesia consultation without cancellation or postponement of surgery

SECONDARY OUTCOMES:
Anesthesia teleconsultation failure rate for technical reasons | up to 1 hour post anesthesia teleconsultation outset
  Rate of patients who did not benefit from anesthesia teleconsultation for technical reasons
Cancellation or postponement surgery rate | 24 hours post surgery
  Patients rate
Patient rate, seen in teleconsultation, secondarily oriented towards a conventional consultation | 24 hours post surgery
  Patients rate
Extension of the ambulatory stay rate | 24 hours post surgery
  Patients rate
Readmitted patients rate | 24 hours post surgery
  Rate of readmitted patients related with surgery and assigned to the teleconsultation
Patient satisfaction with anesthesia teleconsultation | at 7 days post hospital discharge
  Global satisfaction level (regarding the sound and picture quality, respect of confidentiality and privacy, recommend or choose teleconsultation for the next anesthesia consultation) using Numerical Rating Scale from 0 to 10, 0 : extremely unsatisfied, 10= extremely satisfied.
Physician satisfaction with anesthesia teleconsultation | up to 1 hour post anesthesia teleconsultation outset
  Global satisfaction level (regarding the sound and picture quality, respect of confidentiality and privacy, clinical observations collection quality, recommend teleconsultation for the next anesthesia consultation) using Numerical Rating Scale from 0 to 10, 0 : extremely unsatisfied, 10= extremely satisfied.
Cost of transportation from home to hospital | at 7 days post hospital discharge
  Cost ( euros)
Rate of transportation carbon footprint saved using anesthesia teleconsultation | at 7 days post hospital discharge
  co2 equivalent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Applegate RL 2nd, Gildea B, Patchin R, Rook JL, Wolford B, Nyirady J, Dawes TA, Faltys J, Ramsingh DS, Stier G. Telemedicine pre-anesthesia evaluation: a randomized pilot trial. Telemed J E Health. 2013 Mar;19(3):211-6. doi: 10.1089/tmj.2012.0132. Epub 2013 Feb 5. PMID 23384334
- [Background] Charles BL. Telemedicine can lower costs and improve access. Healthc Financ Manage. 2000 Apr;54(4):66-9. PMID 10915354
- [Background] Dilisio RP, Dilisio AJ, Weiner MM. Preoperative virtual screening examination of the airway. J Clin Anesth. 2014 Jun;26(4):315-7. doi: 10.1016/j.jclinane.2013.12.010. Epub 2014 Jun 8. PMID 24916897
- [Background] Galvez JA, Rehman MA. Telemedicine in anesthesia: an update. Curr Opin Anaesthesiol. 2011 Aug;24(4):459-62. doi: 10.1097/ACO.0b013e328348717b. PMID 21659874
- [Background] Huston JL, Burton DC. Patient satisfaction with multispecialty interactive teleconsultations. J Telemed Telecare. 1997;3(4):205-8. doi: 10.1258/1357633971931174. PMID 9614735
- [Background] Wade VA, Karnon J, Elshaug AG, Hiller JE. A systematic review of economic analyses of telehealth services using real time video communication. BMC Health Serv Res. 2010 Aug 10;10:233. doi: 10.1186/1472-6963-10-233. PMID 20696073
- [Background] Wong DT, Kamming D, Salenieks ME, Go K, Kohm C, Chung F. Preadmission anesthesia consultation using telemedicine technology: a pilot study. Anesthesiology. 2004 Jun;100(6):1605-7. doi: 10.1097/00000542-200406000-00038. No abstract available. PMID 15166585